CLINICAL TRIAL: NCT05788055
Title: The Study of Helicobacter Pylori Infection in Acute Myocardial Infarction Patients
Brief Title: Helicobacter Pylori Infection in Acute Myocardial Infarction Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Ezz Mostafa, Dr, Sohag University
Other Study IDs: H.Pylori and AMI
Record Dates: First submitted 2023-03-05; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Coronary Syndrome Patients: Stool Analysis will be done for all cases to detect H.pylori Antigen and results will be analysed into infected patients and non infected patients.
  Interventions: Diagnostic Test: Stool Analysis
- Chronic Stable Angina Patients: Stool Analysis will be done for all cases to detect H.pylori Antigen and results will be analysed into infected patients and non infected patients.
  Interventions: Diagnostic Test: Stool Analysis

INTERVENTIONS:
Diagnostic Test: Stool Analysis — Stool Analysis to detect H.Pylori Antigen in Stool

SUMMARY:
This study aims to investigate the association between H.Pylori and ACS .

DETAILED DESCRIPTION:
The study is based on show the relationship between H.Pylori infection and Acute Coronary Syndrome .

Active H.Pylori infection is common in ACS and may represent a modifiable risk factor for upper gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting by acute coronary syndrome to Coronary Care Units, Internal Medicine Department, Sohag Faculty of Medicine from 18 .

Exclusion Criteria:

* 1.Patients with Cardiogenic Shock. 2. Renal Impairment.(Creatinine Clearence <60) 3. A known systemic inflammatory condition. 4.They had taken any antibiotics in the previous 1 months. 5.They had taken any proton pump inhibitors in previous 2 weeks. 6.Gastrointestinal Bleeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting by acute coronary syndrome to Coronary Care Units and the chronic stable angina patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of results of H.Pylori antigen with ACS | from the day of admission to the day of disharge of sohag university hospitals
  Analysis of H.Pylori antigen and compare with ECG findings and cardiac enzymes

REFERENCES:
- [Background] Lai CY, Yang TY, Lin CL, Kao CH. Helicobacter pylori infection and the risk of acute coronary syndrome: a nationwide retrospective cohort study. Eur J Clin Microbiol Infect Dis. 2015 Jan;34(1):69-74. doi: 10.1007/s10096-014-2207-7. Epub 2014 Jul 26. PMID 25063740